CLINICAL TRIAL: NCT05331950
Title: Predictive and Associated Factors of Musculoskeletal Injuries in Office Workers.
Brief Title: Predictive and Associated Factors of Musculoskeletal Injuries
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Atif Zulfiqar
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Musculoskeletal Injury
Keywords: Functional movement screen.; Musculoskeletal Injury; Office workers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Office workers: The office workers will do their routine job tasks and will be observed through injury predictor (functional movement screen) at baseline and after actual injuries happened 6 months
  Interventions: Other: Office Workers

INTERVENTIONS:
Other: Office Workers — Office Workers which will be observed/exposed with different task and different factors

SUMMARY:
The aim of this research is to find out the factors associated with musculoskeletal injuries among office workers and also determine whether Functional Movement Screen (FMS) can predict musculoskeletal injuries or not? Prospective Cohort study will be done at the offices of Rawalpindi. The sample size is 208. Study duration will be of 6 months. Non probability Purposive Sampling will be used. Tools used in the study are FMS, Fat Caliper, Weighing machine & Inches tape. Data will be analyzed through SPSS 23.

DETAILED DESCRIPTION:
Musculoskeletal injuries and conditions represent a major public health problem, with significant social, economic, and health consequences. Office workers are forming a major group for musculoskeletal injuries as they have to work for a longer period of time on computer and sitting on a chair. Musculoskeletal discomfort in office workers is commonly caused by poor ergonomic workstation design, psychosocial, physical and organizational risk factor. There are several MSK disorders associated with computer use in people spending more than 9 hours or more every day using computer.

To combat workplace caused mental and physical exhaustion physical activity has been proven to be an efficient. Physical activity is known not to only treat but prevent the occurrence of a fore coming disease. Being physically active will lead to reduced stress levels and increased productivity. The Functional Movement Screen (FMS) is a physical examination used to measure essential movement patterns in a practical and dynamic way. Functional Movement screen was designed with a purpose of identify body asymmetries, assess mobility and stability within the kinetic chain of whole-body movements and to detect poor quality movement patterns. Other tools like modified Y-balance test have also been used to predict injuries.

Literature review: Previously in a study carried out on firefighters Contreras et al reported that 47% of the participants had an FMS score lower than 14 and they accounted for 72% of the total musculoskeletal injuries.

In another study carried out on Collegiate athletic association Division II athletes the overall prognostic accuracy of the FMS offered a slightly better than 50/50 chance of correctly classifying those most at risk for injury.

A study carried out to find the association between functional fitness scores calculated by FMS and musculoskeletal injury in police officers by Liana Lentz et al suggested that of all the participants, females accounted for 17.9% of the injured subjects.

Previously a study carried out by Michal Pan Tanowitz et al to find factors associated with musculoskeletal injuries in an infantry commanders' course suggested that army operators who sustained a spinal injury have a significantly greater BMI than those who did not, and also increased body fat combined with reduced physical fitness may increase the soldier's risk for injury.

ELIGIBILITY:
Inclusion Criteria:

* • Both Genders.

  * 25-45 years.
  * Office workers

Exclusion Criteria:

* any neuromusculoskeletal injuries

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: office workers spending at least 6 hours per day at work
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen | 1 day
  The assessment of Functional movement screen is based on qualitative analysis with a four-point ranking system (From 0 to 3). To evaluate movement quality, 3-performs the movement correctly without any compensation, complying with standard movement expectations associated with each test; 2-able to complete the movement but must compensate in some way to perform the fundamental movement; 1-unable to complete the movement pattern or is unable to assume the position to perform the movement; 0-pain anywhere in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- MTBC, Rawalpindi, Punjab Province, Pakistan